CLINICAL TRIAL: NCT03663309
Title: Assessment of Adherence to Gluten Free Diet in Children and Adolescents by Detection of Gluten Immunogenic Peptides in Faecal Samples and Nutritional Assessment. Retrospective Study
Brief Title: Assessment of Adherence to Gluten Free Diet in Children and Adolescents by Detection of Gluten in Faecal Samples.
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, raanan shamir, Professor, Rabin Medical Center
Other Study IDs: 0367-17RMC
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Celiac Disease in Children
MeSH Terms: interventions — Defecation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: 1. Children and adolescents aged 2-17 years, reported to be on gluten free diet for at least a year, diagnosed with celiac disease
  2. Children and adolescents aged 2-17 years that are reported to be noncompliant with gluten free diet, diagnosed with celiac disease for at least 1 year.
  Interventions: Diagnostic Test: detecting Gluten peptides in faecal and urine samples
- control group: Healthy controls aged 2-17 years old matched for age and sex.

INTERVENTIONS:
Diagnostic Test: detecting Gluten peptides in faecal and urine samples — At each visit patient will:
  * Bring 4-day food diary (attached)
  * Fill symptoms and complaints questionnaire (attached)
  * Provide 24 h diet recall in case a food diary absents
  * Fill Biagi score questionnaire (attached)
  * Perform blood test of TTG
  * Provide stool and urine samples
  Groups: study group

SUMMARY:
To assess the adherence to gluten free diet by measuring faecal and urinary gluten immunogenic peptides (GIP). This will provide an objective measure for adherence.

DETAILED DESCRIPTION:
The adherence to the GFD can be assessed through a dietary interview performed by a registered dietitian or patient self-reports, mucosal healing, assessed by a small bowel biopsy or CD serological screening tests showing decreasing levels of antibodies. However, none of these methods offer an accurate measure of dietary compliance. A novel method to monitor the adherence to the GFD by detection of immune-dominant gluten peptides in human faeces or urine using the anti-α -gliadin G12 antibody was described recently in the literature. Gluten peptides, in particular peptides equivalent to the immunogenic - α -gliadin-33-mer peptide, are resistant to gastrointestinal digestion and that ensures a significant amount of the ingested gluten is excreted in faeces. Consequently, recovery of detectable amounts of the immunogenic fraction in faeces or urine indicates that gluten has passed through the digestive tract, and in the case of urine was absorbed, and, therefore, that gluten has been consumed .

ELIGIBILITY:
Inclusion Criteria:

* Age 2-17 years.
* Either diagnosis of celiac disease or, in controls, no systemic disease or inflammation
* For all groups parents will provide informed consent.

Exclusion Criteria:

° Children with suspected or known inflammatory bowel disease or other gastrointestinal or systemic diseases.

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: 1. Children and adolescents aged 2-17 years, reported to be on gluten free diet for at least a year, diagnosed with celiac disease
  2. Children and adolescents aged 2-17 years that are reported to be noncompliant with gluten free diet, diagnosed with celiac disease for at least 1 year.
  3. Healthy controls aged 2-17 years old matched for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Correlation between fecal gluten peptides and nutritional assessment for gluten free diet, and correlation with celiac serology. | one year
  Our goal is to examine which method will be the most accurate, nutritional assessment or laboratory tests for the adherence to GFD

CONTACTS AND LOCATIONS:
Overall Officials: Liron Mondshine, B.Sc, Study Chair — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided